CLINICAL TRIAL: NCT03800511
Title: Prediction of Intra-abdominal Adhesion Before CS: A Diagnostic Test Study
Brief Title: Prediction of Intra-abdominal Adhesion Before CS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nahed allam (Other)
Responsible Party: Sponsor-Investigator, Nahed allam, Proffesor Nahed Ezzat Allam (Nallam, Al-Azhar University
Organization: Al-Azhar University (Other)
Other Study IDs: Prediction of intra-abdominal
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Intra-Abdominal; Adhesion
Keywords: sliding test , ceaserean section
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- repeated caesarean section: full term pregnant women with singleton baby with a history of at least previous one caesarean section
  Interventions: Diagnostic Test: sliding test

INTERVENTIONS:
Diagnostic Test: sliding test — ultrasound detected sliding test before doing repeated caesarean section
  Other Names: ultrasound detected sliding test

SUMMARY:
Recognition of intraabdominal adhesion before doing repeated cesarean section is helpful for the surgeon and patients.

DETAILED DESCRIPTION:
the repeated cesarean section is associated with recorded maternal morbidity including placenta preavia and accreta , liability to injuries to the bladder, intestine or vascular injuries. The anticipation of the problem is important for decreasing its adverse effect . preoperative diagnosis of pelvic adhesion between the uterus and anterior abdominal wall, bladder, intestine or omentum could b of help to give time for a surgeon to prepare senior staff obstetrician or others and theatre requirements to overcome any problem happened.

ELIGIBILITY:
Inclusion Criteria:

* pregnant in their 9th-month singleton, planned for elective CS and had a history of previous CS

Exclusion Criteria:

* included multiple pregnancies, preterm labour, emergency CS, skin burn at the site of CS

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women in their 9th-month singleton planned for elective repeated CS and had a history of previous CS
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
intra-abdominal adhesion | intra-operative period
  presence of adhesion between uterus and abdominal wall or intestine on bladder

SECONDARY OUTCOMES:
skin to uterine incision time | intra-operative period
  time consumed by surgeon from skin incision to uterine incision in minutes
need to insert intra-peritoneal drain | intraoperative period
  if there in marked adhesion and vascular injury a drain could be inserted

CONTACTS AND LOCATIONS:
Overall Officials: Taiseer Maarouf, MD, Study Chair — Al-Azhar University

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.discussion with the other authors after completion of recruitment of patients